CLINICAL TRIAL: NCT05262972
Title: APPLICATION OF ULTRASOUND-GUIDED PERCUTANEOUS ELECTROLYSIS IN THE PAIN OF THE SECOND METATARSOPHALANGEAL JOINT IN ADULT WOMEN
Brief Title: Percutaneous Needle Electrolysis on Metatarsalgia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Blanca de la Cruz Torres, Director, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PNE and metatarsalgia
Record Dates: First submitted 2022-02-19; First posted 2022-03-02 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Metatarsalgia
MeSH Terms: conditions — Metatarsalgia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental): The subject will obtain a conservative treatment for this type of pathology consisting of the development of a personalized plantar orthosis
  Interventions: Other: Conservatory treatment
- Group II (Experimental): The subjects belonging to this group, in addition to providing their corresponding personalized plantar orthosis, will receive a complementary treatment consisting of the application of ultrasound-guided percutaneous electrolysis
  Interventions: Other: Innovate treatment

INTERVENTIONS:
Other: Conservatory treatment — Personalized plantar orthosis
  Arms: Group I
Other: Innovate treatment — Personalized plantar orthosis + percutaneous electrolysis
  Arms: Group II

SUMMARY:
Percutaneous electrolysis is a minimally invasive method that involves the application of a galvanic current through an acupuncture needle. The needle is placed directly into the soft tissue structures, essential with ultrasound guidance. This technique involves the combination of mechanical stimulation produced by the needle and electrical/biochemical stimulation provided by the electrical current.

Endogenous pain modulation shows clinical relevance of this technique and plays an important role in the experience of pain.

Plantar plate injury is a pathology that frequently occurs in the forefoot, especially in middle-aged women, causing metatarsalgia that is sometimes very intense. In most cases it is secondary to a mechanical imbalance of the forefoot, related to an insufficiency of the first radius. For this reason, the researchers hypothesize that the application of ultrasound-guided percutaneous electrolysis on the plantar plate, combined with the conservative treatment consisting of the development of a personalized plantar orthosis, can cause positive effects in the patient's clinic as well as improve their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Adult female patients (40-65 years old)
* Having pain in the 2nd MTP joint of the foot due to pathology of the plantar plate, diagnosed by a specialized professional.

Exclusion Criteria:

* to have suffered an injury to their musculoskeletal system in the last 6 months.
* to have the present neuritic pathology,
* to have complete rupture of the plantar plate, 2nd finger supraadductus, flexor digitorum longus tenosynovitis,
* to have problems in the lumbar spine,
* to have undergone surgery in the lumbar spine or lower limbs.
* to use a plantar orthosis.
* to have the presence of associated pathologies in the foot,
* to be under the influence of any medication at the time of the study, fear of needles
* to be pregnant
* to be epileptic.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — This pathology is much more frequent in women.
Enrollment: 30 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Quality of life | 1 month
  Foot Health Status Questionnaire
Subjetive level of pain | 1 month
  Intensity of subjective pain in the injured structure (0, no pain; 10, worse pain)
level of pain at palpation | 1 month
  Intensity of pain on palpation in the injured structure (0, no pain; 10, worse pain)
Distribution of plantar pressures | 1 month
  Podiatric platform (pressure percentage 0-100%)

CONTACTS AND LOCATIONS:
Locations (1):
- Blanca de la Cruz, Seville, Spain